CLINICAL TRIAL: NCT06179186
Title: Hair Removal by Intense Pulsed Light Versus Diode Laser: Randomized Controlled Clinical Trial
Brief Title: Hair Removal: Intense Pulsed Light Versus Diode Laser
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early after interim analysis of 48 participants, which showed significant group differences with 80% power, making further enrollment unnecessary.
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Christiane Pavani, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTBB
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hair Removal
Keywords: hair removal; diode laser; photoepilation; intense pulsed light; epilation; Depilation
MeSH Terms: interventions — Intense Pulsed Light Therapy; Random Allocation; Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: Participants are assigned two groups in parallel for the duration of the study
Who Masked: Participant, Outcomes Assessor
Masking Description: participants will receive both treatments in right and left axilla, and they won´t know which treatment will be performed at each side.
  The outcome assessor won´t know which treatment was performed at the axilla.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intense Pulsed Light (Experimental): The hair from axilla of one side of the body will be removed with 4 sessions of Intense Pulsed Light
  Interventions: Device: Intense Pulsed Light; Device: Diode Laser
- Diode laser (Experimental): The hair from axilla of one side of the body will be removed with 4 sessions of Diode Laser
  Interventions: Device: Intense Pulsed Light; Device: Diode Laser

INTERVENTIONS:
Device: Intense Pulsed Light — The axilla will be treated with intense pulsed light, being right or left, depending upon randomization.
  Other Names: Randomized
Device: Diode Laser — The axilla will be treated with diode laser, being right or left, depending upon randomization.
  Other Names: Randomized

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of two hair removal techniques: Intense Pulsed Light (IPL) and Diode Laser in woman underarm. .

Main Questions:

* Determine the thread count in a 4cm² quadrant in the central axillary region before each session, 4-6 weeks after the last session and at follow-up 30 weeks after the last session;
* Measure the thickness of the hair before each session, 4-6 weeks after the last session and at follow-up 6 months after the last session;
* Compare the level of pain during procedures;
* Evaluate the volunteer's level of satisfaction after the end of the sessions programmed by the study;
* Evaluate quality of life and self-image before and after the end of the sessions programmed by the study;
* Evaluate the maintenance of results 6 months after the last procedure performed.

Researchers will compare IPL and Diode laser to see if hair removal is similar at short and long time course.

The IPL treatment will be applied to one axilla. The 800nm Diode Laser treatment will be applied to the other axilla. Treatment allocation will be randomized for each participant. Participants will undergo monthly sessions for four months, totaling four treatments. Follow-up assessments will occur 30 days and 6 months after the final session.

DETAILED DESCRIPTION:
This is a randomized controlled trial of hair removal in axilla for women, being intense pulsed light compared to diode laser.

The session frequency will be once a month for 4 months, totaling 4 treatments. There will be a follow-up at 30 days and 6 months after the end of the treatment.

After the evaluations and photographs, the armpits will be cleaned with 0.5% alcoholic chlorhexidine and will be shaved with a disposable razor blade. Neutral water-based gel will be applied to the region to receive the treatment. Patients will be instructed not to perform any trichotomy procedures in the region during the research period.

The treatment technique will be punctual where the applicator will be kept in full contact with the skin at 90° and moved to the next point after deposition of energy over the entire treatment area until the defined energy is delivered. The applicator tip will be cooled as much as the equipment allows.

ELIGIBILITY:
Inclusion Criteria:

* Female patients,
* aged 18 and older,
* with a complaint of hair in the axillary region,
* Fitzpatrick skin phototype I to IV,
* presenting dark hair

Exclusion Criteria:

* Patients who have used medications that alter hair production,
* Patients who have used medications that are photosensitizing,
* Patients who have used isotretinoin or vitamin A-synthesized acids, antibiotics such as tetracycline,
* Patients using anticoagulant
* Patients with vitiligo or epilepsy,
* Pregnant or lactating individuals,
* those with active herpes,
* Patient with history of tumors,
* Patient with axillary scarring (hyper or hypotrophic),
* Patient who have used another method of hair removal involving complete hair removal by pulling with a minimum period of 30 days from the date of the initial assessment, or have used another laser hair removal method in the treatment area,
* Immunocompromised patients,
* Patients with sun-sensitive skin with inflammation,
* Individuals with psoriasis,
* Patients with tattoos on the application site,
* Patients who have undergone ovary removal or have reached menopause

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Hair count | before each session (S0,Month1, Month2, Month3), 4-6 weeks after the last session (Month4) and at follow-up 24 weeks after the last session (Month 10).
  The counting of the hairs will be performed by observing the visible hairs in the treatment area photographs of the volunteers. In this way, a percentage comparison will be made in relation to the initial number of hairs. The hair count will be conducted in a 4cm² quadrant in the central axillary region.
Global Aesthetic Improvement Scale (GAIS) | 4-6 weeks after the last session (Month4) and at follow-up 24 weeks after the last session (Month 10).
  The photographs will be evaluated by two independent and blind evaluators, making a comparison between the photos before the procedure (S0) and the final effect of the short-term (S4) and long-term (S5) treatment. The evaluations will be classified according to the percentage of change: no results 0% reduction, bad reduction 0% to 25%, average 25% to 50%, good 50% to 75% and excellent 75%-100%.

SECONDARY OUTCOMES:
Hair Thickness | before each session (S0,Month1, Month2, Month3), 4-6 weeks after the last session (Month4) and at follow-up 24 weeks after the last session (Month 10).
  Images of the demarcated region will be obtained using a dermatoscope (5 images per region per assessment). The hair thickness will be measured using the Image J software (NIH).
Pain Score (Visual Analogue Scale) | before each session (S0,Month1, Month2, Month3), 4-6 weeks after the last session (Month4) and at follow-up 24 weeks after the last session (Month 10).
  Immediately after the end of the procedure in each armpit, the patient will respond using the visual analogue scale (VAS) to the sensation of pain perceived during the procedure.
  It consists of a straight line, 10 centimeters long, where one end represents the total absence of pain and the other end represents the most intense pain possible. The person experiencing the pain is asked to mark a point on the line that represents the intensity of the pain they are experiencing. The marked point can be measured in centimeters from the end that represents the absence of pain.
Quality of Live | before first session (S0), and at follow-up 24 weeks after the last session (Month 10).
  The WHOQOL-bref quality of life questionnaire consists of 26 questions, with responses following a Likert scale (from 1 to 5, with higher scores indicating better quality of life) his questionnaire includes 2 questions that assess overall quality of life, while the remaining questions make up 4 domains (physical, psychological, social relationships, and environment).
Satisfaction level Score | At follow-up 24 weeks after the last session (Month 10).
  The patient's satisfaction level with the treatment will be assessed through a questionnaire containing five multiple-choice questions. These questions will address the degree of discomfort experienced during the sessions, how many sessions this discomfort persisted, the satisfaction level regarding the achieved results, the perceived percentage improvement in the concern, and, finally, how likely the patient would recommend the undergone treatment to someone with a similar concern. Each response receive 1 up to 5 points, and the total Score varies from 4 to 20, being the highest as the highest the satisfaction.
Self - Esteem Scale | before first session (S0) and at follow-up 24 weeks after the last session (Month 10).
  The Self - Esteem Rosenberg Scale consists of 10 statements related to self-evaluation and self-acceptance. Respondents must indicate their level of agreement or disagreement with each statement on a response scale that typically ranges from "strongly disagree" to "strongly agree." The statements are mostly positive and are used to assess the extent to which a person feels positive or negative about themselves.

OTHER OUTCOMES:
Adverse events | before each session (S0,Month1, Month2, Month3), 4-6 weeks after the last session (Month4) and at follow-up 24 weeks after the last session (Month 10).
  Adverse effects noted during and after treatments will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Pavani, PhD, Study Director — University of Nove de Julho
Locations (2):
- Brazil (2):
  - Universidade Nove de Julho, São Paulo, São Paulo
  - Ambulatório Universidade Nove de Julho, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No